CLINICAL TRIAL: NCT03750097
Title: Validation of a Commercially Available Smartwatch for Step Detection in Persons With Multiple Sclerosis
Brief Title: Validation of a Smartwatch in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Neurological Rehabilitation Center Quellenhof (Unknown); ZTM Bad Kissingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ms-bewegt-Validation
Record Dates: First submitted 2018-07-30; First posted 2018-11-21 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Motion sensors; Smartwatch; Steps; Walking; Validation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking protocol (Experimental): Walking for 250 steps with comfortable walking velocity (CWV), slow walking velocity (SWV: CWV - 20%) and fast walking velocity (FWV: CWV + 20%) with sufficient rest between conditions.
  Interventions: Behavioral: Comfortable walking velocity (CWV); Behavioral: Slow walking velocity (SWV: CWV - 20%); Behavioral: Fast walking velocity (FWV: CWV + 20%)

INTERVENTIONS:
Behavioral: Comfortable walking velocity (CWV) — Walking for 250 Steps with self-selected comfortable walking velocity while wearing the two accelerometers (Polar M600 and ActiGraph wGT3X-BT)
Behavioral: Slow walking velocity (SWV: CWV - 20%) — Walking for 250 Steps with slow walking velocity while wearing the two accelerometers (Polar M600 and ActiGraph wGT3X-BT). Slow walking consists of walking with 20% slower than the self-selected comfortable walking velocity by following a researcher who controls the walking velocity with a measuring wheel.
Behavioral: Fast walking velocity (FWV: CWV + 20%) — Walking for 250 Steps with fast walking velocity while wearing the two accelerometers (Polar M600 and ActiGraph wGT3X-BT). Fast walking consists of walking with 20% faster than the self-selected comfortable walking velocity by following a researcher who controls the walking velocity with a measuring wheel.

SUMMARY:
The study is designed to validate the accuracy of steps detected by a commercially available smartwatch in persons with multiple sclerosis. Specifically, the investigators examine whether a smartwatch can detect steps accurately during slow, comfortable and fast overground walking. The total steps counted by the smartwatch will be compared to those counted by an accelerometer commonly used in clinical studies and the actually walked steps.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system. It is one of the most common neurological diseases in young adulthood. The main symptoms of MS are gait and mobility impairments, which also determine the severity of the disease. Currently, subjective clinical functional tests are commonly used to evaluate therapy outcomes. Due to advancing mechanization, body-worn accelerometers have been established as a potential instrument for the objective detection of mobility in clinical research. The accuracy of these devices for determining the mobility is therefore essential. However, current studies, especially in people with altered gait, show large deviations in step detection accuracy.

In the present study we want to investigate: i) whether a commercially available smartwatch (Polar M600) counts steps in persons with multiple sclerosis (pwMS) accurately and ii) whether it counts steps as accurately as an accelerometer commonly used in clinical research (ActiGraph wGT3X-BT). In addition, the accuracy of the step detection by the algorithms of the manufacturer of the two devices (Polar M600 and ActiGraph wGT3X-BT) will be compared with an own-developed algorithm.

For this purpose, 63 pwMS with low to severe functional restriction (EDSS: 0 - 6.5) will participate in this validation study. The validation protocol consists of three walking tests with different walking velocities. During these three conditions the participants will wear the Polar M600 on the wrist and the ActiGraph wGT3X-BT with a belt over the hip. In the first walking test, the subjects will complete 250 steps with comfortable walking velocity (CWV). After a sufficient break, the participants will be randomly assigned to either a fast walking velocity condition (FWV: CWV + 20%) followed by a sufficient period of rest and a slow walking velocity condition (SWV: CWV - 20%) or vice versa. Each of the walking tests with modified walking velocity also consists of 250 steps. To analyze the accuracy of step detection, the measured steps of the devices will be compared with the actually walked 250 steps.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis with Expanded Disability Status Scale between 0 - 6.5
* Ability to walk 250 steps with or without an assistive device

Exclusion Criteria:

* Clinically relevant cardiovascular or orthopaedic disease
* Severe polyneuropathy
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Step detection during comfortable walking | Following the comfortable walking velocity protocol, an average of 2 minutes
  Step detection accuracy of the two devices (Polar M600 and ActiGraph wGT3X-BT) for both the standard algorithm and the self-developed algorithm during comfortable walking for 250 steps.

SECONDARY OUTCOMES:
Step detection during slow walking | Following the slow walking velocity protocol, an average of 2 minutes
  Step detection accuracy of the two devices (Polar M600 and ActiGraph wGT3X-BT) for both the standard algorithm and the self-developed algorithm during slow walking for 250 steps.
Step detection during fast walking | Following the fast walking velocity protocol, an average of 2 minutes
  Step detection accuracy of the two devices (Polar M600 and ActiGraph wGT3X-BT) for both the standard algorithm and the self-developed algorithm during fast walking for 250 steps.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Department of Sport Science and Sport; Peter Flachenecker, Prof. Dr. med., Principal Investigator — Neurological Rehabilitation Center Quellenhof
Locations (1):
- Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Department of Sport Science and Sport, Gebbertstr. 123b, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Project webpage — http://www.sport.fau.de/ms-bewegt/